CLINICAL TRIAL: NCT01575600
Title: Effect of Intravenous Fluid Therapy on Postoperative Vomiting in Children Undergoing Otorhinolaryngological Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ignacio Cortínez F. (Other)
Responsible Party: Sponsor-Investigator, Ignacio Cortínez F., Profesor Asociado, Departamento de Anestesiología, Pontificia Universidad Catolica de Chile
Organization: Pontificia Universidad Catolica de Chile (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 10-095
Record Dates: First submitted 2012-04-10; First posted 2012-04-11 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Postoperative Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 10 mL/kg/h lactated Ringer's solution (Active Comparator): Group 1, 10 mL/kg/h lactated Ringer's solution
  Interventions: Other: Intraoperative lactated Ringer's solution
- 30 mL/kg/h lactated Ringer's solution (Experimental): Group 2, 30 mL/kg/h lactated Ringer's solution
  Interventions: Other: Intraoperative lactated Ringer's solution

INTERVENTIONS:
Other: Intraoperative lactated Ringer's solution — After induction, IV access was established and children were randomly allocated to receive one of two interventions: Group 1, 10 mL/kg/h lactated Ringer's solution; Group 2, 30 mL/kg/h lactated Ringer's solution.

SUMMARY:
The purpose of this randomized clinical trial is to evaluate the interaction of intravenous fluid therapy during otorhinolaryngological surgery, on postoperative vomiting. The hypothesis is that perioperative supplemental intravenous fluid administration reduces the incidence of postoperative vomiting.

DETAILED DESCRIPTION:
Postoperative vomiting is a common complication on pediatric surgery, especially otorhinolaryngological surgery. Is one of the main reasons of prolonged hospital stay, and also a cause of patient´s discomfort and an increase on hospitalization cost.

There are studies in adults with inconclusive results related to supplemental fluid therapy and decrease of postoperative nausea and vomiting. But, in recent years a study in children showed favorable results in strabismus surgery. The foundation of this study consist in that hypovolemia may possibly cause a decrease in perfusion causing intestinal hypoxia, which in turn increase the incidence of nausea and vomiting. The objective of this study is to observe the effect of supplemental fluid therapy on postoperative vomiting on otorhinolaryngological surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I or II
* Age 1-12 yr
* Scheduled for elective tonsillectomy or adenotonsillectomy

Exclusion Criteria:

* History of diabetes
* History of mental retardation
* Obesity (BMI ≥95th percentile for age and sex)
* Intake of antiemetic or psychoactive medication within 24 hours before surgery
* Known gastroesophageal reflux

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2010-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Vomiting at 24 hours postoperative | First 24 hours postoperative
  Presence of at least one episode of vomiting in the first 24 hours postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinico Universidad Catolica, Santiago, Santiago Metropolitan, Chile